CLINICAL TRIAL: NCT05465317
Title: Comparative Cardiovascular and Renal Effectiveness and Safety of Empagliflozin and Other SGLT2i in Patients With Type 2 Diabetes (T2D) With and Without Baseline Kidney Disease in the United States
Brief Title: Evaluating Comparative Effectiveness of Empagliflozin in Type 2 Diabetes Population With and Without Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0228
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Empagliflozin initiators: Patient with type 2 diabetes, with or without Chronic Kidney Disease (CKD), who initiated Empagliflozin between January 1, 2016 and December 31, 2020.
  Interventions: Drug: Empagliflozin
- Dipeptidyl peptidate-4 inhibitor (DPP4i) initiators: Patient with type 2 diabetes, with or without Chronic Kidney Disease (CKD), who initiated dipeptidyl peptidate-4 inhibitor (DPP4i) between January 1, 2016 and December 31, 2020.
  Interventions: Drug: Dipeptidyl Peptidate-4 inhibitors

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin
  Groups: Empagliflozin initiators
Drug: Dipeptidyl Peptidate-4 inhibitors — Dipeptidyl Peptidate-4 inhibitors
  Groups: Dipeptidyl peptidate-4 inhibitor (DPP4i) initiators

SUMMARY:
The primary purpose of this research study is to determine the cardiovascular and renal effectiveness and safety of empagliflozin compared to dipeptidyl peptidase-4 inhibitors (DPP4i) in patients with Type 2 Diabetes Mellitus (T2DM) with and without established kidney disease.

The secondary purpose of this research study is to determine the cardiovascular and renal effectiveness and safety of any Sodium glucose co-transporter-2 inhibitors (SGLT2i) compared to Glucagon-like Peptide-1 Receptor Agonists (GLP1RA) in patients with T2DM.

ELIGIBILITY:
Inclusion criteria:

* Patients ≥18 years old
* Having a diagnosis of type 2 diabetes in 12 months before the index date (defined as the date of initiation of empagliflozin or Glucagon-like Peptide-1 Receptor Agonists (GLP1RA) or Dipeptidyl Peptidate-4 inhibitor (DPP4i), based on the cohort evaluated), based on International Classification of Diseases (ICD)-9 and -10 codes and other available data
* Record of prescription for empagliflozin, any Sodium glucose co-transporter-2 inhibitors (SGLT2i), any DPP4 inhibitor, or any GLP1RA use between 1 January 2015 and 31 December 2020, and
* No record of any prescription for the drugs being compared during the 12 months + 30-day grace preceding the index date period, i.e.,

  * For the primary comparison of initiation of empagliflozin versus DPP4i, patients will not have any prescription for empagliflozin/any SGLT2i or DPP4i during the preceding 12 months + 30-day grace period.
  * For the comparison of initiation of SGLT2i versus GLP1RA, patients will not have any prescription for SGLT2i or GLP1RA during the preceding 12 months + 30-day grace period.
  * For the comparison of initiation of empagliflozin versus GLP1RA, patients will not have any prescription for empagliflozin/any SGLT2i or GLP1RA during the preceding 12 months + 30-day grace period.

Exclusion criteria:

* Aged <18 years on the first prescription date of the qualifying prescription,
* Pre-existing diagnosis of type 1 diabetes mellitus (T1DM) during the 12 months before the index date,
* Having a disqualifying diagnosis during the 12 months before the index date, defined as having at least one of the following: estimated glomerular filtration rate (eGFR) <30, dialysis, polycystic kidney disease or a kidney transplant,
* <12 months of available data before the index date, and/or no complete history of drug dispensations/other records of drug use during this period, defined as not having at least 1 ambulatory visit and at least 1 medication prescription during the preceding 12 months, and
* Missing or ambiguous data on serum creatinine in the 12 months prior to the index date or sex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The analysis will include adults (≥18 years) with type 2 diabetes with or without kidney disease in the US.
Sampling Method: Non-Probability Sample
Enrollment: 62197 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Edmonston D, Mulder H, Lydon E, Chiswell K, Lampron Z, Shay C, Marsolo K, Shah RC, Jones WS, Gordon H, Hwang W, Ayoub I, Ford D, Chamberlain A, Rao A, Fonseca V, Chang A, Ahmad F, Hung A, Hunt K, Butler J, Bosworth HB, Pagidipati N. Kidney and Cardiovascular Effectiveness of SGLT2 Inhibitors vs GLP-1 Receptor Agonists in Type 2 Diabetes. J Am Coll Cardiol. 2024 Aug 20;84(8):696-708. doi: 10.1016/j.jacc.2024.06.016. PMID 39142723
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional, retrospective cohort study (NIS) using existing data from 20 US health systems, the study period was from 1 Jan 2014 through 31 December 2021, to determine the cardiovascular and renal effectiveness and safety up to 24 months after initiation of empagliflozin compared to dipeptidyl peptidate-4 inhibitor (DPP4i) in patients with type 2 diabetes.
Pre-assignment Details: Only subjects that met all the study inclusion and none of the exclusion criteria were to be entered in the study.
Period: Overall Study
Arm/Group | Empagliflozin Initiators | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators
Started | 20279 | 41918
Completed | 20279 | 41918
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Primary study cohort: Patient with type 2 diabetes who initiated Empagliflozin or Dipeptidyl peptidate-4 inhibitor (DPP4i) between January 1, 2016 and December 31, 2020. Based on existing data from 20 United States (US) health systems that have mapped their electronic health record (EHR) data to the National Patient-Centered Clinical Research Network (PCORnet) Common Data Model.
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin Initiators | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators | Total
Number analyzed (Participants) | 20279 | 41918 | 62197
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60.0 [52.0 to 67.0] | 63.0 [54.0 to 72.0] | 62.0 [53.0 to 70.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9551 | 22007 | 31558
  Male | 10728 | 19911 | 30639
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15006 | 29510 | 44516
  Black | 4198 | 9641 | 13839
  Other | 1075 | 2767 | 3842

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of the Composite Outcome Including 40% Decline in Estimated Glomerular Filtration Rate (eGFR), Incident End-stage Renal Disease (ESRD) and All-cause Death
Description: 40% decline in eGFR: at least 2 measurements during follow-up of at least a 40% decline relative to baseline separated by >= 28 days. the second eGFR measurement is required to be within 2 years from index, at which time, all patients were censored.
  ESKD: at least 1 kidney transplant or ESKD diagnosis/procedure or at least 2 dialysis diagnoses/procedures separated by >= 28 days or eGFR<15 on 2 measurements separated by >= 28 days.
  Post-LASSO overlap weighting was used. A LASSO penalized regression model was created with covariates of interest, subgroup variables, and all pairwise interactions. Variables chosen by the LASSO model were refit to a logistic model in order to calculate the PS estimates. The overlap weights were then created such that the weights were equal to the PS for participants prescribed the reference treatment (DPP4i) and 1-PS for participants prescribed empagliflozin.
  Results are presented for the overall cohort and for the CKD and non-CKD cohorts.
Time Frame: Starting the day after the index date (date of initiation of empagliflozin or DPP4i) and continuing until the first occurrence of the outcome of interest, or end of study date (date of death, date of study end, 2 years after index date). Up to 2 years.
Population: as for baseline characteristics
Measure: Number; unit: (First) events per 1000 patient years
Groups:
- Empagliflozin Initiators - Propensity Scored-weighted: Patient with type 2 diabetes, with or without Chronic Kidney Disease (CKD), who initiated Empagliflozin between January 1, 2016 and December 31, 2020. The cohort was propensity scored-weighted.
- Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted: Patient with type 2 diabetes, with or without Chronic Kidney Disease (CKD), who initiated dipeptidyl peptidate-4 inhibitor (DPP4i) between January 1, 2016 and December 31, 2020. The cohort was propensity scored-weighted.
- Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort: Patient with type 2 diabetes, with established Chronic Kidney Disease (CKD), who initiated Empagliflozin between January 1, 2016 and December 31, 2020. The cohort was propensity scored-weighted.
- DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort: Patient with type 2 diabetes with established Chronic Kidney Disease (CKD), who initiated dipeptidyl peptidate-4 inhibitor (DPP4i) between January 1, 2016 and December 31, 2020. The cohort was propensity scored-weighted.
- Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort: Patient with type 2 diabetes, without established Chronic Kidney Disease (CKD), who initiated Empagliflozin between January 1, 2016 and December 31, 2020. The cohort was propensity scored-weighted.
- DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort: Patient with type 2 diabetes without established Chronic Kidney Disease (CKD), who initiated dipeptidyl peptidate-4 inhibitor (DPP4i) between January 1, 2016 and December 31, 2020. The cohort was propensity scored-weighted.
Arm/Group | Empagliflozin Initiators - Propensity Scored-weighted | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted | Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort | DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort | Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort | DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort
Number analyzed (Participants) | 20279 | 41918 | 3633 | 11126 | 16646 | 30792
(First) events per 1000 patient years | 26.65 | 36.65 | 44.15 | 67.36 | 22.62 | 29.33
Statistical Analysis 1: Comparison: Empagliflozin Initiators - Propensity Scored-weighted vs Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted; Outcomes were assessed using Cox proportional hazards (PH) models in a 2-arm comparison. The analysis included all patients with a valid overlap weight and was performed using the reweighted population. The main analysis assessed outcomes while patients remain on initial treatment; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.65 to 0.86] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 2: Comparison: Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort vs DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.001, Regression, Cox; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.52 to 0.86] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 3: Comparison: Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort vs DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.008, Regression, Cox; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.67 to 0.94] — Ratio calculated as Empagliflozin/DPP4i

2. Secondary Outcome: Incidence Rate of the 40% Decline in Estimated Glomerular Filtration Rate (eGFR)
Description: 40% decline in eGFR: at least 2 measurements (second measurement must be within 2 years) during follow-up of at least a 40% decline relative to baseline separated by >= 28 days.
  Post-LASSO (least absolute shrinkage and selection operator) overlap weighting was used. A LASSO penalized regression model was created with the covariates of interest, subgroup variables, and all pairwise covariate-subgroup interactions. Outcome for this model was treatment group (DPP4i as the reference). The variables chosen by the LASSO model were refit to a logistic model in order to calculate the propensity score (PS) estimates. The overlap weights were then created such that the weights were equal to the PS for participants prescribed the reference treatment (DPP4i) and 1-PS for participants prescribed empagliflozin.
  Results are presented for the overall cohort and separately for the CKD and non-CKD cohorts.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: (First) events per 1000 patient years
Arm/Group | Empagliflozin Initiators - Propensity Scored-weighted | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted | Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort | DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort | Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort | DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort
Number analyzed (Participants) | 20279 | 41918 | 3633 | 11126 | 16646 | 30792
(First) events per 1000 patient years | 12.10 | 16.55 | 16.46 | 27.39 | 11.10 | 13.95
Statistical Analysis 1: Comparison: Empagliflozin Initiators - Propensity Scored-weighted vs Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.005, Regression, Cox; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.60 to 0.91] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 2: Comparison: Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort vs DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.02, Regression, Cox; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.41 to 0.91] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 3: Comparison: Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort vs DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.08, Regression, Cox; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.63 to 1.03] — Ratio calculated as Empagliflozin/DPP4i

3. Secondary Outcome: Incidence Rate of End-stage Kidney Disease (ESKD)
Description: ESKD definition: at least 1 kidney transplant or ESKD diagnosis/procedure or at least 2 dialysis diagnoses/procedures separated by >= 28 days or eGFR<15 on 2 measurements separated by >= 28 days.
  Post-LASSO (least absolute shrinkage and selection operator) overlap weighting was used. A LASSO penalized regression model was created with the covariates of interest, subgroup variables, and all pairwise covariate-subgroup interactions. Outcome for this model was treatment group (DPP4i as the reference). The variables chosen by the LASSO model were refit to a logistic model in order to calculate the propensity score (PS) estimates. The overlap weights were then created such that the weights were equal to the PS for participants prescribed the reference treatment (DPP4i) and 1-PS for participants prescribed empagliflozin.
  Results are presented for the overall cohort and separately for the CKD and non-CKD cohorts.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: (First) events per 1000 patient years
Arm/Group | Empagliflozin Initiators - Propensity Scored-weighted | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted | Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort | DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort | Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort | DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort
Number analyzed (Participants) | 20279 | 41918 | 3633 | 11126 | 16646 | 30792
(First) events per 1000 patient years | 3.34 | 4.90 | 8.18 | 12.96 | 2.23 | 2.97
Statistical Analysis 1: Comparison: Empagliflozin Initiators - Propensity Scored-weighted vs Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.05, Regression, Cox; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.46 to 1.00] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 2: Comparison: Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort vs DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.09, Regression, Cox; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.35 to 1.09] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 3: Comparison: Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort vs DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.30, Regression, Cox; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.43 to 1.29] — Ratio calculated as Empagliflozin/DPP4i

4. Secondary Outcome: Incidence Rate of Dialysis
Description: Incident dialysis, given dialysis in the 12 months preceding index date is a disqualifying diagnosis/procedure.
  Post-LASSO (least absolute shrinkage and selection operator) overlap weighting was used. A LASSO penalized regression model was created with the covariates of interest, subgroup variables, and all pairwise covariate-subgroup interactions. Outcome for this model was treatment group (DPP4i as the reference). The variables chosen by the LASSO model were refit to a logistic model in order to calculate the propensity score (PS) estimates. The overlap weights were then created such that the weights were equal to the PS for participants prescribed the reference treatment (DPP4i) and 1-PS for participants prescribed empagliflozin.
  Results are presented for the overall cohort and separately for the CKD and non-CKD cohorts.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: (First) events per 1000 patient years
Arm/Group | Empagliflozin Initiators - Propensity Scored-weighted | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted | Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort | DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort | Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort | DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort
Number analyzed (Participants) | 20279 | 41918 | 3633 | 11126 | 16646 | 30792
(First) events per 1000 patient years | 3.47 | 4.76 | 7.86 | 12.03 | 2.46 | 3.01
Statistical Analysis 1: Comparison: Empagliflozin Initiators - Propensity Scored-weighted vs Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.11, Regression, Cox; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.49 to 1.08] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 2: Comparison: Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort vs DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.12, Regression, Cox; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.35 to 1.12] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 3: Comparison: Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort vs DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.52, Regression, Cox; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.50 to 1.42] — Ratio calculated as Empagliflozin/DPP4i

5. Secondary Outcome: Incidence Rate of Kidney Transplant
Description: Kidney transplant: any procedure associated with healthcare encounters, including hospitalizations and specialist outpatient and primary care encounters.
  Post-LASSO (least absolute shrinkage and selection operator) overlap weighting was used. A LASSO penalized regression model was created with the covariates of interest, subgroup variables, and all pairwise covariate-subgroup interactions. Outcome for this model was treatment group (DPP4i as the reference). The variables chosen by the LASSO model were refit to a logistic model in order to calculate the propensity score (PS) estimates. The overlap weights were then created such that the weights were equal to the PS for participants prescribed the reference treatment (DPP4i) and 1-PS for participants prescribed empagliflozin.
  Results are presented for the overall cohort and separately for the CKD and non-CKD cohorts.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: (First) events per 1000 patient years
Arm/Group | Empagliflozin Initiators - Propensity Scored-weighted | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted | Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort | DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort | Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort | DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort
Number analyzed (Participants) | 20279 | 41918 | 3633 | 11126 | 16646 | 30792
(First) events per 1000 patient years | 0.02 | 0.06 | 0.10 | 0.10 | 0.00 | 0.05

6. Secondary Outcome: Incidence Rate of Composite Outcome Including Acute Hospitalization for Heart Failure and All-cause Death
Description: Composite outcome including acute hospitalization for heart failure and All-cause death: Any diagnosis of heart failure associated with hospital admission, including inpatient and emergency department (ED) to inpatient encounters. From death records provided by sites, supplemented with linkage using Datavant Software.
  Post-LASSO overlap weighting was used. A LASSO penalized regression model was created with covariates of interest, subgroup variables, and all pairwise interactions. Variables chosen by the LASSO model were refit to a logistic model in order to calculate the PS estimates. The overlap weights were then created such that the weights were equal to the PS for participants prescribed the reference treatment (DPP4i) and 1-PS for participants prescribed empagliflozin.
  Results are presented for the overall cohort and separately for the CKD and non-CKD cohorts.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: (First) events per 1000 patient years
Arm/Group | Empagliflozin Initiators - Propensity Scored-weighted | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted | Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort | DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort | Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort | DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort
Number analyzed (Participants) | 20279 | 41918 | 3633 | 11126 | 16646 | 30792
(First) events per 1000 patient years | 24.65 | 30.24 | 50.05 | 61.34 | 18.86 | 22.83
Statistical Analysis 1: Comparison: Empagliflozin Initiators - Propensity Scored-weighted vs Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.02, Regression, Cox; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.72 to 0.97] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 2: Comparison: Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort vs DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.12, Regression, Cox; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.65 to 1.05] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 3: Comparison: Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort vs DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.10, Regression, Cox; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.70 to 1.03] — Ratio calculated as Empagliflozin/DPP4i

7. Secondary Outcome: Incidence Rate of Acute Hospitalization for Heart Failure
Description: Acute hospitalization for heart failure: Any diagnosis of heart failure associated with hospital admission, including inpatient and emergency department (ED) to inpatient encounters.
  Post-LASSO (least absolute shrinkage and selection operator) overlap weighting was used. A LASSO penalized regression model was created with the covariates of interest, subgroup variables, and all pairwise covariate-subgroup interactions. Outcome for this model was treatment group (DPP4i as the reference). The variables chosen by the LASSO model were refit to a logistic model in order to calculate the propensity score (PS) estimates. The overlap weights were then created such that the weights were equal to the PS for participants prescribed the reference treatment (DPP4i) and 1-PS for participants prescribed empagliflozin.
  Results are presented for the overall cohort and separately for the CKD and non-CKD cohorts.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: (First) events per 1000 patient years
Arm/Group | Empagliflozin Initiators - Propensity Scored-weighted | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted | Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort | DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort | Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort | DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort
Number analyzed (Participants) | 20279 | 41918 | 3633 | 11126 | 16646 | 30792
(First) events per 1000 patient years | 12.74 | 14.40 | 29.47 | 33.08 | 8.92 | 9.95
Statistical Analysis 1: Comparison: Empagliflozin Initiators - Propensity Scored-weighted vs Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.32, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.72 to 1.11] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 2: Comparison: Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort vs DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.50, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.65 to 1.24] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 3: Comparison: Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort vs DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.50, Regression, Cox; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.68 to 1.20] — Ratio calculated as Empagliflozin/DPP4i

8. Secondary Outcome: Incidence Rate of All-cause Death
Description: All-cause death, from death records provided by sites, supplemented with linkage using Datavant Software.
  Post-LASSO (least absolute shrinkage and selection operator) overlap weighting was used. a LASSO penalized regression model was created with the covariates of interest, subgroup variables, and all pairwise covariate-subgroup interactions. Outcome for this model was treatment group (DPP4i as the reference). The variables chosen by the LASSO model were refit to a logistic model in order to calculate the propensity score (PS) estimates. The overlap weights were then created such that the weights were equal to the PS for participants prescribed the reference treatment (DPP4i) and 1-PS for participants prescribed empagliflozin.
  Results are presented for the overall cohort and separately for the CKD and non-CKD cohorts.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: (First) events per 1000 patient years
Arm/Group | Empagliflozin Initiators - Propensity Scored-weighted | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted | Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort | DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort | Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort | DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort
Number analyzed (Participants) | 20279 | 41918 | 3633 | 11126 | 16646 | 30792
(First) events per 1000 patient years | 13.47 | 18.60 | 23.75 | 35.56 | 11.09 | 14.49
Statistical Analysis 1: Comparison: Empagliflozin Initiators - Propensity Scored-weighted vs Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.005, Regression, Cox; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.62 to 0.92] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 2: Comparison: Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort vs DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.03, Regression, Cox; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.49 to 0.96] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 3: Comparison: Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort vs DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.074, Regression, Cox; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.63 to 1.02] — Ratio calculated as Empagliflozin/DPP4i

9. Secondary Outcome: Incidence Rate of the Composite Outcome Including MI, Stroke, All-cause Death and Coronary Revascularization Procedure
Description: Composite outcome including MI, Stroke, All-cause death and Coronary revascularization procedure: For MI and stroke, any inpatient diagnosis associated with healthcare encounters, including inpatient and ED to inpatient For all-cause death, death records provided by sites, supplemented with linkage using Datavant Software.
  Post-LASSO overlap weighting was used. A LASSO penalized regression model was created with covariates of interest, subgroup variables, and all pairwise interactions. Variables chosen by the LASSO model were refit to a logistic model in order to calculate the PS estimates. The overlap weights were then created such that the weights were equal to the PS for participants prescribed the reference treatment (DPP4i) and 1-PS for participants prescribed empagliflozin.
  Results are presented for the overall cohort and separately for the CKD and non-CKD cohorts.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: (First) events per 1000 patient years
Arm/Group | Empagliflozin Initiators - Propensity Scored-weighted | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted | Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort | DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort | Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort | DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort
Number analyzed (Participants) | 20279 | 41918 | 3633 | 11126 | 16646 | 30792
(First) events per 1000 patient years | 97.31 | 96.36 | 169.32 | 164.13 | 81.63 | 80.89
Statistical Analysis 1: Comparison: Empagliflozin Initiators - Propensity Scored-weighted vs Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.46, Regression, Cox; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.95 to 1.12] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 2: Comparison: Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort vs DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.63, Regression, Cox; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.90 to 1.20] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 3: Comparison: Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort vs DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.52, Regression, Cox; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.94 to 1.14] — Ratio calculated as Empagliflozin/DPP4i

10. Secondary Outcome: Incidence Rate of the Composite Outcome Including MI, Stroke, All-cause Death (MACE)
Description: Composite outcome including MI, Stroke, All-cause death: For MI and stroke, any inpatient diagnosis associated with healthcare encounters, including inpatient and ED to inpatient For all-cause death, death records provided by sites, supplemented with linkage using Datavant Software.
  Post-LASSO overlap weighting was used. A LASSO penalized regression model was created with covariates of interest, subgroup variables, and all pairwise interactions. Variables chosen by the LASSO model were refit to a logistic model in order to calculate the PS estimates. The overlap weights were then created such that the weights were equal to the PS for participants prescribed the reference treatment (DPP4i) and 1-PS for participants prescribed empagliflozin.
  Results are presented for the overall cohort and separately for the CKD and non-CKD cohorts.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: (First) events per 1000 patient years
Arm/Group | Empagliflozin Initiators - Propensity Scored-weighted | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted | Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort | DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort | Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort | DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort
Number analyzed (Participants) | 20279 | 41918 | 3633 | 11126 | 16646 | 30792
(First) events per 1000 patient years | 23.93 | 30.27 | 40.65 | 55.67 | 20.07 | 24.18
Statistical Analysis 1: Comparison: Empagliflozin Initiators - Propensity Scored-weighted vs Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.007, Regression, Cox; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.70 to 0.94] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 2: Comparison: Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort vs DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.03, Regression, Cox; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.57 to 0.97] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 3: Comparison: Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort vs DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.10, Regression, Cox; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.71 to 1.03] — Ratio calculated as Empagliflozin/DPP4i

11. Secondary Outcome: Incidence Rate of Diabetic Ketoacidosis
Description: Any diabetic ketoacidosis diagnosis associated with healthcare encounters in the inpatient setting.
  Post-LASSO (least absolute shrinkage and selection operator) overlap weighting was used. A LASSO penalized regression model was created with the covariates of interest, subgroup variables, and all pairwise covariate-subgroup interactions. Outcome for this model was treatment group (DPP4i as the reference). The variables chosen by the LASSO model were refit to a logistic model in order to calculate the propensity score (PS) estimates. The overlap weights were then created such that the weights were equal to the PS for participants prescribed the reference treatment (DPP4i) and 1-PS for participants prescribed empagliflozin.
  Results are presented for the overall cohort and separately for the CKD and non-CKD cohorts.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: (First) events per 1000 patient years
Groups:
- Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort: Patient with type 2 diabetes, with established kidney disease, who initiated Empagliflozin between January 1, 2016 and December 31, 2020. The cohort was propensity scored-weighted.
Arm/Group | Empagliflozin Initiators - Propensity Scored-weighted | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted | Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort | DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort | Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort | DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort
Number analyzed (Participants) | 20279 | 41918 | 3633 | 11126 | 16646 | 30792
(First) events per 1000 patient years | 4.06 | 2.86 | 3.59 | 3.46 | 4.17 | 2.71
Statistical Analysis 1: Comparison: Empagliflozin Initiators - Propensity Scored-weighted vs Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.15, Regression, Cox; Hazard Ratio (HR) = 1.37, 95% CI 2-sided [0.89 to 2.10] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 2: Comparison: Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort vs DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.93, Regression, Cox; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.40 to 2.72] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 3: Comparison: Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort vs DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.113, Regression, Cox; Hazard Ratio (HR) = 1.47, 95% CI 2-sided [0.91 to 2.38] — Ratio calculated as Empagliflozin/DPP4i

12. Secondary Outcome: Incidence Rate of Severe Hypoglycemia
Description: Any severe hypoglycemia diagnosis associated with healthcare encounters in the inpatient or ED setting.
  Post-LASSO (least absolute shrinkage and selection operator) overlap weighting was used. A LASSO penalized regression model was created with the covariates of interest, subgroup variables, and all pairwise covariate-subgroup interactions. Outcome for this model was treatment group (DPP4i as the reference). The variables chosen by the LASSO model were refit to a logistic model in order to calculate the propensity score (PS) estimates. The overlap weights were then created such that the weights were equal to the PS for participants prescribed the reference treatment (DPP4i) and 1-PS for participants prescribed empagliflozin.
  Results are presented for the overall cohort and separately for the CKD and non-CKD cohorts.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: (First) events per 1000 patient years
Arm/Group | Empagliflozin Initiators - Propensity Scored-weighted | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted | Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort | DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort | Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort | DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort
Number analyzed (Participants) | 20279 | 41918 | 3633 | 11126 | 16646 | 30792
(First) events per 1000 patient years | 9.43 | 10.69 | 14.90 | 18.89 | 8.17 | 8.72
Statistical Analysis 1: Comparison: Empagliflozin Initiators - Propensity Scored-weighted vs Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.43, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.71 to 1.16] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 2: Comparison: Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort vs DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.32, Regression, Cox; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.51 to 1.24] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 3: Comparison: Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort vs DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.81, Regression, Cox; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.71 to 1.30] — Ratio calculated as Empagliflozin/DPP4i

13. Secondary Outcome: Incidence Rate of Urinary Tract Cancer
Description: Two or more urinary tract cancer diagnoses associated with healthcare encounters within 2 months.
  Post-LASSO (least absolute shrinkage and selection operator) overlap weighting was used. A LASSO penalized regression model was created with the covariates of interest, subgroup variables, and all pairwise covariate-subgroup interactions. Outcome for this model was treatment group (DPP4i as the reference). The variables chosen by the LASSO model were refit to a logistic model in order to calculate the propensity score (PS) estimates. The overlap weights were then created such that the weights were equal to the PS for participants prescribed the reference treatment (DPP4i) and 1-PS for participants prescribed empagliflozin.
  Results are presented for the overall cohort and separately for the CKD and non-CKD cohorts.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: (First) events per 1000 patient years
Arm/Group | Empagliflozin Initiators - Propensity Scored-weighted | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted | Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort | DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort | Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort | DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort
Number analyzed (Participants) | 20279 | 41918 | 3633 | 11126 | 16646 | 30792
(First) events per 1000 patient years | 4.65 | 5.14 | 8.62 | 9.35 | 3.74 | 4.13
Statistical Analysis 1: Comparison: Empagliflozin Initiators - Propensity Scored-weighted vs Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.69, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.65 to 1.33] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 2: Comparison: Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort vs DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.82, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.51 to 1.70] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 3: Comparison: Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort vs DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.76, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.60 to 1.45] — Ratio calculated as Empagliflozin/DPP4i

14. Secondary Outcome: Incidence Rate of Severe Urinary Tract Infections (UTI)
Description: Any severe Urinary Tract Infections (UTI) diagnosis associated with healthcare encounters in the inpatient or ED setting for Pyelonephritis or Urosepsis.
  Post-LASSO (least absolute shrinkage and selection operator) overlap weighting was used. A LASSO penalized regression model was created with the covariates of interest, subgroup variables, and all pairwise covariate-subgroup interactions. Outcome for this model was treatment group (DPP4i as the reference). The variables chosen by the LASSO model were refit to a logistic model in order to calculate the propensity score (PS) estimates. The overlap weights were then created such that the weights were equal to the PS for participants prescribed the reference treatment (DPP4i) and 1-PS for participants prescribed empagliflozin.
  Results are presented for the overall cohort and separately for the CKD and non-CKD cohorts.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: (First) events per 1000 patient years
Arm/Group | Empagliflozin Initiators - Propensity Scored-weighted | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted | Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort | DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort | Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort | DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort
Number analyzed (Participants) | 20279 | 41918 | 3633 | 11126 | 16646 | 30792
(First) events per 1000 patient years | 0.69 | 1.01 | 0.90 | 2.00 | 0.64 | 0.77
Statistical Analysis 1: Comparison: Empagliflozin Initiators - Propensity Scored-weighted vs Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.39, Regression, Cox; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.29 to 1.62] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 2: Comparison: Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort vs DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.34, Regression, Cox; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.09 to 2.27] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 3: Comparison: Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort vs DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.72, Regression, Cox; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.29 to 2.33] — Ratio calculated as Empagliflozin/DPP4i

15. Secondary Outcome: Incidence Rate of Acute Kidney Injury (AKI) That Requires Dialysis
Description: Any Acute kidney injury diagnosis associated with inpatient healthcare encounters for AKI plus at least one inpatient encounter indicating dialysis within 28 days of the AKI encounter. Two or more dialysis encounters separated by 28 days or more was excluded from this definition.
  Post-LASSO overlap weighting was used. A LASSO penalized regression model was created with covariates of interest, subgroup variables, and all pairwise interactions. Variables chosen by the LASSO model were refit to a logistic model in order to calculate the PS estimates. The overlap weights were then created such that the weights were equal to the PS for participants prescribed the reference treatment (DPP4i) and 1-PS for participants prescribed empagliflozin.
  Results are presented for the overall cohort and separately for the CKD and non-CKD cohorts.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: (First) events per 1000 patient years
Arm/Group | Empagliflozin Initiators - Propensity Scored-weighted | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted | Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort | DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort | Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort | DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort
Number analyzed (Participants) | 20279 | 41918 | 3633 | 11126 | 16646 | 30792
(First) events per 1000 patient years | 1.23 | 1.45 | 2.53 | 4.02 | 0.93 | 0.83
Statistical Analysis 1: Comparison: Empagliflozin Initiators - Propensity Scored-weighted vs Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.62, Regression, Cox; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.43 to 1.66] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 2: Comparison: Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort vs DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.31, Regression, Cox; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.21 to 1.64] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 3: Comparison: Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort vs DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.76, Regression, Cox; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.46 to 2.92] — Ratio calculated as Empagliflozin/DPP4i

16. Secondary Outcome: Incidence Rate of Genital Mycotic Infection
Description: Any genital mycotic infection diagnosis associated with healthcare encounters, including hospitalizations and outpatient encounters, or prescription for fluconazole.
  Post-LASSO (least absolute shrinkage and selection operator) overlap weighting was used. A LASSO penalized regression model was created with the covariates of interest, subgroup variables, and all pairwise covariate-subgroup interactions. Outcome for this model was treatment group (DPP4i as the reference). The variables chosen by the LASSO model were refit to a logistic model in order to calculate the propensity score (PS) estimates. The overlap weights were then created such that the weights were equal to the PS for participants prescribed the reference treatment (DPP4i) and 1-PS for participants prescribed empagliflozin.
  Results are presented for the overall cohort and separately for the CKD and non-CKD cohorts.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: (First) events per 1000 patient years
Arm/Group | Empagliflozin Initiators - Propensity Scored-weighted | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted | Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort | DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort | Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort | DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort
Number analyzed (Participants) | 20279 | 41918 | 3633 | 11126 | 16646 | 30792
(First) events per 1000 patient years | 115.96 | 65.32 | 99.20 | 52.23 | 119.94 | 68.52
Statistical Analysis 1: Comparison: Empagliflozin Initiators - Propensity Scored-weighted vs Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators - Propensity Scored-weighted; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 1.72, 95% CI 2-sided [1.58 to 1.88] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 2: Comparison: Empagliflozin Initiators - Chronic Kidney Disease (CKD) Cohort vs DPP4i Initiators - Chronic Kidney Disease (CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 1.84, 95% CI 2-sided [1.48 to 2.30] — Ratio calculated as Empagliflozin/DPP4i
Statistical Analysis 3: Comparison: Empagliflozin Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort vs DPP4i Initiators - Non-Chronic Kidney Disease (Non-CKD) Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 1.70, 95% CI 2-sided [1.54 to 1.87] — Ratio calculated as Empagliflozin/DPP4i

ADVERSE EVENTS:
Time Frame: Starting the day after the index date (date of initiation of empagliflozin or DPP4i) and continuing until the first occurrence of the outcome of interest, or end of study date (date of death, date of study end, 2 years after index date). Up to 2 years.
Description: No adverse events (AEs) were collected on an individual case level. Serious AEs and Other AEs are not collected in the database. All-Cause Mortality is an outcome of this study and thus additionally reported below.
  Patient with type 2 diabetes who initiated Empagliflozin or Dipeptidyl peptidate-4 inhibitor (DPP4i) between January 1, 2016 and December 31, 2020. Based on existing data from 20 US health systems that have mapped their EHR data to the National PCORnet Common Data Model.
Arm/Group | Empagliflozin Initiators | Dipeptidyl Peptidate-4 Inhibitor (DPP4i) Initiators
All-Cause Mortality (participants affected / at risk) | 341/20279 | 1528/41918
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Limitations inherent to all electronic health record (EHR) based studies, including potential for missing data (i.e., data that was generated through a different health system) or inaccurate data based on billing codes. This limitation could have resulted in HCRU not captured in the current study which could have attenuated the observed results (e.g., medications, hospitalizations, etc).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT05465317/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT05465317/SAP_001.pdf